CLINICAL TRIAL: NCT04740112
Title: Effects of Beta-glucan and Product Claims for Breakfast Bars on Appetite Response and Consumer Preference: a Randomized Controlled Trial
Brief Title: Beta-glucan, Product Claims and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2021/01/7
Record Dates: First submitted 2021-01-27; First posted 2021-02-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Food

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control breakfast bar with low dietary fiber without product claims (Placebo Comparator)
  Interventions: Other: Foods with beta-glucan from oats and barley
- Test breakfast bar with high dietary fiber without product claims (Experimental)
  Interventions: Other: Foods with beta-glucan from oats and barley
- Test breakfast bar with high dietary fiber with product claims (Experimental)
  Interventions: Other: Foods with beta-glucan from oats and barley

INTERVENTIONS:
Other: Foods with beta-glucan from oats and barley — Breakfast bars made with varying levels of total dietary fiber and beta-glucan, with or without claims on package image
  Other Names: Food

SUMMARY:
This is a digital clinical trial to investigate satiety and consumer preference in responses to three test breakfast bars with varying level of dietary fiber, beta-glucan, and product packages (with or without product claims) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-70 years.
* Habitual snack bar consumers (consume bars at least 3 times a week).
* Body mass index 20-29.9 kg/m² (based on self-reported weight and height).
* Understand the study procedures.
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Willing to follow study procedures on test days.
* Willing to abstain from strenuous exercise, consuming alcoholic drinks 24 hours before the test day.
* Willing to provide informed consent to participate in the study.
* Willing to maintain confidentiality of the study and test products.

Exclusion Criteria:

* Pregnant or lactating women, or women who are planning to become pregnant during the study
* Known food allergies, sensitivity, or intolerance to any food or food ingredients
* Participating in another clinical trial for food, investigational drug, nutritional supplement, or lifestyle modification
* Taking medications that affect appetite, metabolism, or blood pressure
* Taking supplements with dietary fiber
* Presence of acute diseases or infection
* Presence or history of chronic diseases
* Diagnosed with eating disorders
* Restraint eaters
* Lost or gained 5 pounds or more in the past 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Hunger | 30 minutes after consumption
  Hunger as measured by visual analog scales in mm using appetite questionnaires
Hunger | 60 minutes after consumption
  Hunger as measured by visual analog scales in mm using appetite questionnaires
Hunger | 90 minutes after consumption
  Hunger as measured by visual analog scales in mm using appetite questionnaires
Hunger | 120 minutes after consumption
  Hunger as measured by visual analog scales in mm using appetite questionnaires
Hunger | 180 minutes after consumption
  Hunger as measured by visual analog scales in mm using appetite questionnaires
Fullness | 30 minutes after consumption
  Fullness as measured by visual analog scales in mm using appetite questionnaires
Fullness | 60 minutes after consumption
  Fullness as measured by visual analog scales in mm using appetite questionnaires
Fullness | 90 minutes after consumption
  Fullness as measured by visual analog scales in mm using appetite questionnaires
Fullness | 120 minutes after consumption
  Fullness as measured by visual analog scales in mm using appetite questionnaires
Fullness | 180 minutes after consumption
  Fullness as measured by visual analog scales in mm using appetite questionnaires
Desire to eat | 30 minutes after test meal consumption
  Desire to eat as measured by visual analog scales in mm using appetite questionnaires
Desire to eat | 60 minutes after test meal consumption
  Desire to eat as measured by visual analog scales in mm using appetite questionnaires
Desire to eat | 90 minutes after test meal consumption
  Desire to eat as measured by visual analog scales in mm using appetite questionnaires
Desire to eat | 120 minutes after test meal consumption
  Desire to eat as measured by visual analog scales in mm using appetite questionnaires
Desire to eat | 180 minutes after test meal consumption
  Desire to eat as measured by visual analog scales in mm using appetite questionnaires
Prospective consumption | 30 minutes after test meal consumption
  Prospective consumption as measured by visual analog scales in mm using appetite questionnaires
Prospective consumption | 60 minutes after test meal consumption
  Prospective consumption as measured by visual analog scales in mm using appetite questionnaires
Prospective consumption | 90 minutes after test meal consumption
  Prospective consumption as measured by visual analog scales in mm using appetite questionnaires
Prospective consumption | 120 minutes after test meal consumption
  Prospective consumption as measured by visual analog scales in mm using appetite questionnaires
Prospective consumption | 180 minutes after test meal consumption
  Prospective consumption as measured by visual analog scales in mm using appetite questionnaires

SECONDARY OUTCOMES:
Flavor rating | 30 minutes after test meal consumption
  Subjective ratings on liking of the product flavor using Likert scales
Sweetness rating | 30 minutes after test meal consumption
  Subjective ratings on sweetness of the product using Likert scales
Texture rating | 30 minutes after test meal consumption
  Subjective ratings on liking of the product texture using Likert scales
Overall product liking | 30 minutes after test meal consumption
  Subjective ratings on overall liking of the product using Likert scales
Purchase intent | 180 minutes after test meal consumption
  Likelihood of buying the product using Likert scales

CONTACTS AND LOCATIONS:
Locations (1):
- No physical visit to a research facility is required., Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No